CLINICAL TRIAL: NCT00198159
Title: A Phase II Study of ZD1839 (Iressa)in Chemotherapy Refractory Germ Cell Tumors Expressing Epidermal Growth Factor Receptor (EGFR)
Brief Title: A Phase II Study of Iressa in Patients With Chemo Refractory Germ Cell Tumors Expressing EGFR
Acronym: IUCRO-0021
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: AstraZeneca (Industry)
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0211-07
Record Dates: First submitted 2005-09-08; First posted 2005-09-20 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Refractory Germ Cell Tumors Expressing EGRF
Keywords: Refractory Germ Cell Tumors; Germ Cell Tumors
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Gefitinib

INTERVENTIONS:
Drug: ZD1839 Iressa

SUMMARY:
This study will evaluate the use of ZD1839 in the treatment of subjects with refractory germ cell tumors. Subjects will take ZD1839 for one year in the absence of excessive toxicity or decision to withdraw.

DETAILED DESCRIPTION:
The primary objective is to determine the response rate of ZD1839 in patients with refractory germ cell tumors expressing EGFR. The secondary objectives are to determine the duration of response, time to progression and overall survival in patients with refractory germ cell tumors expressing EGFR and treated with ZD1839; to evaluate the tolerability of ZD1839 in patients with refractory germ cell tumors and to correlate tumor response to degree of EGFR expression by immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or serologic proof of metastatic germ cell neoplasm(gonadal or extragonadal primary) with disease not amenable to cure with either surgery or chemotherapy. Patients w/ seminoma and non-seminoma are eligible, as are women w/ ovarian germ cell tumors.
* Evidence of recurrent or metastatic carcinoma
* Must have received initial cisplatin combination therapy & demonstrated progression following the administration of at least one "salvage" regimen for advanced germ cell neoplasms.
* Patients are eligible after first line platinum bsed chemotherapy if their disease has relapsed and they have primary mediastinal non seminomatous germ cell tumor, late relapse or progressed w/in 4 wks of last platinum dose.
* immunohistochemical documentation of EGFR expression documented.
* adequate organ function: ANC >/=150,plt >100K, total bili </= upper limit of normal(ULN). Pts w/ liver mets up to 3x ULN.Transaminases up to 1.5 x ULN if alk phos is </=ULN or alk phos may be up to 4x ULN if transaminases are </= ULN. Pts w/ liver mets may have alk phos up to 5x ULN. Serum crt </= 2.0.
* ECOG performance status 0-2.

Exclusion Criteria:

* Must be 3 weeks post major surgery, radiotherapy, or chemotherapy and hae recovered from all toxicity.
* Active unresolved infection and/or are receiving concurrent treatment with parenteral antibiotics are ineligible.
* Patients requiring steroids for symptomatic brain metastasis are not eligible.
* Pregnant or lactating patients are not eligible.
* Class III/IV heart disease

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21
Dates: Start 2002-09; Primary Completion 2006-02 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To determine the response rate of ZD1839

SECONDARY OUTCOMES:
To determine duration of response, time to progression and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Einhorn, M, Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States